CLINICAL TRIAL: NCT03477617
Title: A Single Centre Feasibility Randomized Controlled Trial of Advanced Minimally Invasive Monitoring to Optimize Hemodynamic Management in Major Noncardiac Surgery
Brief Title: Advanced Monitoring to Inform and Guide Perioperative Hemodynamic Optimization 1 (AMIGO-1) Study
Acronym: AMIGO-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Jo Carroll, Principal Investigator, University Health Network, Toronto
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 15-9764
Record Dates: First submitted 2018-02-26; First posted 2018-03-26 (Actual); Last update posted 2020-09-29 (Actual); Status verified 2020-09

CONDITIONS: Intraoperative Fluid Management

STUDY DESIGN:
Intervention Model Description: Parallel Assignment Participants are randomized to two groups; both groups will have an intraoperative minimally invasive cardiac output monitor connected.
  In the intervention arm, the anesthesiologist will treat episodes of hypotension using a hemodynamic algorithm based on the information for the cardiac output monitor.
  In the control arm, the anesthesiologist will treat episodes of hypotension using standard of care management and will be blinded to the information from the cardiac output monitor. Data from the monitor will be stored for comparison between the arms.
  This is a pilot study; therefore, the main objective is to assess feasibility of a future multicenter RCT, based on the following domains: (i) participation rate among eligible patients; (ii) practicality of implementing the study intervention in a clinical setting; (iii) collect descriptive data for differences between the 2 arms; (iv) collect safety data to ensure no harm has resulted from the study protocol
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intraoperative Hemodynamic Algorithm (Experimental): In the experimental group, the anesthesiologist will have complete access to data from the minimal invasive cardiac output monitor. During the intraoperative period, the anesthesiologist will be instructed to use a hemodynamic management algorithm to manage episodes of significant hypotension
  Interventions: Other: Intraoperative Hemodynamic Algorithm
- Usual Hemodynamic Management (Active Comparator): In the control arm, the participant will be monitored by the cardiac output monitor, but the anesthesiologists in the operating room will be blinded to hemodynamic data from the monitor. Data from the monitor will be stored electronically and used to compare hemodynamic parameters between study arms.
  Interventions: Combination Product: Usual hemodynamic management

INTERVENTIONS:
Other: Intraoperative Hemodynamic Algorithm — Anesthesiologists are instructed to use the study's algorithm to manage intraoperative hypotension in response to the cardiac output monitor values.
  Arms: Intraoperative Hemodynamic Algorithm
Combination Product: Usual hemodynamic management — Anesthesiologists are instructed to manage intraoperative hypotension based on their usual clinical care, without information from cardiac output monitor
  Arms: Usual Hemodynamic Management

SUMMARY:
Serious complications occur in about 16% of major surgeries. Episode of hypotension during surgery may be a leading cause of these complications. Even though hypotension occurs frequently during surgery, choosing the correct treatment remains difficult in clinical practice. Physicians are often uncertain as to whether low blood pressure should be treated with intravenous fluid or vasoactive drugs. The first treatment of choice typically involves administering more intravenous fluid; however, excessive fluid administration during surgery has been shown to be deleterious. New minimally invasive hemodynamic monitors now offer a potential solution by guiding physicians with respect to the choice of appropriate intervention (i.e., fluid versus vasoactive drugs). The Investigators will conduct a single-center feasibility randomized control trial (RCT) at the Toronto General Hospital (Toronto, ON, Canada) of an algorithm to manage hypotension during surgery based on the information captured by a minimally invasive monitor. Sixty participants who are aged 40 years or older and scheduled to undergo an abdominal, pelvic or vascular surgery will be randomized to have the intraoperative hypotension managed by either the new algorithm (guided by the monitor) or usual care. Participants will be recruited over 12 to 18 months, and followed for 30 days to describe differences in clinical care, hemodynamics, complications, and death. The feasibility of a future multicenter RCT will be assessed based on this present study demonstrating that (1) the algorithm can be practically implemented in a clinical setting where hemodynamic monitors are not typically used; (2) initial descriptive data suggest differences in care between groups; (3) there are no obvious major harms from the protocol; and (4) there is an acceptable participation rate among eligible patients. These data will inform any required changes to the algorithm and protocol to allow for its application in a future study.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥40 years
* Abdominal, retroperitoneal, pelvic or vascular surgery requiring general anesthesia and planned postoperative stay of ≥48 hours for medical reasons
* Elevated perioperative cardiovascular risk based on at least one of the following:

  * cardiovascular comorbidities: coronary artery disease, heart failure, cerebrovascular disease, or peripheral arterial disease
  * elevated age (≥70 y),
  * smoker,
  * hypertension,
  * diabetes mellitus,
  * or preoperative estimated glomerular filtration rate ≤60mL/min/1.73m2
* Planned placement of invasive arterial line for clinical care

Exclusion Criteria:

* Preoperative dialysis dependence
* Minimally invasive procedures (i.e., laparoscopic or endovascular approach)
* Intra-thoracic procedures
* Non-sinus rhythm
* Liver resection surgery

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-05-03 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
Survey score on practicality of study algorithm (Intervention) | 2 years
  • Practicality of study algorithm will be measured by the survey scores of the anesthesiologists involved in the intraoperative care, assessing several domains using a 5 point Likert scale such as (1) Ease of use, (2) Clinical Utility, (3) Validity
Participation rate (Feasibility trial pre-RCT) | 2 years
  • Participation rate: The number of patients consented to the study over the number of eligible patients. This will help estimate recruitment rates in a future clinical randomized trial.
Incidence of treatment related Adverse Events | 2 years
  Number of participants with Adverse Events thought to be at least possibly related to the study treatment will be reported. This outcome will assure that no harm has resulted from the study protocol and the protocol is safe for a future randomized control trial

SECONDARY OUTCOMES:
Volume of intravenous fluid and volume of blood products (therapeutic interventions) for each arm of the study. | During intra-operative period and recovery, an average of 12 hours.
  • The volume of IV fluid and volume of blood products prescribed by the anesthesiologist will be reported as mean (in mL) separately for each study arm. Since this is a feasibility trial the statistical analysis for this study will be descriptive in nature, therefore no statistical differences will be reported between the 2 arms.
Dose of vasoactive medication (therapeutic interventions) for each arm of the study. | During intra-operative period and recovery, an average of 12 hours.
  • The dose of vasoactive medications prescribed by the anesthesiologist will be reported as means (in the unit of each vasoactive medication i.e., mg, mcg, etc.) separately for each study arm. Since this is a feasibility trial the statistical analysis for this study will be descriptive in nature, therefore no statistical differences will be reported between the 2 arms.
Hypotension (blood pressure in mmHg) (therapeutic interventions) for each arm of the study | During intra-operative period and up to 72 hours after surgery.
  • Hypotension is the indication for receiving treatment in the study; therefore, blood pressure will be measured during surgery (every 5 minutes electronically by the non-invasive monitors) and after surgery (every hour by an ambulatory blood pressure monitor) separately for each study arm. Since this is a feasibility trial the statistical analysis for this study will be descriptive in nature, therefore no statistical differences will be reported between the 2 arms.

CONTACTS AND LOCATIONS:
Overall Officials: Duminda N Wijeysundera, Dr, Principal Investigator — Universtiy Health Network. Toronto General Hospital
Locations (1):
- Toronto General Hospital, University Health Network, Toronto, Ontario, Canada